CLINICAL TRIAL: NCT06935279
Title: Ultrastructural Pathology and Pathophysiology of Atherosclerotic Plague With Intracellular Bactria
Brief Title: Types of Intracellular Bacteria in Atherosclerotic Plaques and Analysis of Risk Factors
Acronym: TiBacAP
Status: Recruiting | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Bei Liu Tangdu; 202501-03 (Other Grant/Funding Number: IEC of Institution for National Drug Clinical Trials, Tangdu Hospital, Fourth Military Medical University)
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Carotid Artery Stenosis; Carotid Artery Stenosis Asymptomatic; Carotid Artery Stenosis Symptomatic; Cerebral Infarction; Transient Ischemic Attack (TIA); Hypertension and Cardiovascular Risk Factors; Hypertension, Essential; Diabetes; Hyperlipidemia
Keywords: atherosclerosis; intracellular bacteria; Carotid plaque
MeSH Terms: conditions — Carotid Stenosis; Cerebral Infarction; Ischemic Attack, Transient; Hypertension; Essential Hypertension; Diabetes Mellitus; Hyperlipidemias; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Carotid Endarterectomy (CEA) is a surgical procedure to reconstruct the carotid arteries by removing atherosclerotic plaque from within the carotid arteries in order to eliminate the source of intracranial embolic foci and improve blood flow. The procedure is usually indicated for patients with moderate carotid stenosis with symptoms or severe carotid stenosis. The clinical samples for this study were all from carotid plaques removed by CEA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- xi'an/Tangdu hospital
  Interventions: Procedure: Head and neck vascular recanalization

INTERVENTIONS:
Procedure: Head and neck vascular recanalization — Head and neck vascular recanalization

SUMMARY:
The goal of this iBacAP study is to identify the types of carotid plaques containing intracellular bacteria in patients with atherosclerosis and to look for associated risk factors. The main questions it aims to answer are the type and distribution of intracellular bacteria in patients' plaques, and whether patients with different intracellular bacterial species have a worse prognosis.

The researchers will comparatively analyse the presence of intracellular bacteria in the plaques of patients with different types of carotid artery stenosis and how diverse they are, and observe whether the type of intracellular bacteria has an impact on prognosis.

Participants will:

1. all participants will have no intervention, conventional treatment including conditioning and surgery.

DETAILED DESCRIPTION:
Main research objectives This project foresees the establishment of a registry of patients and specimen banks after carotid endarterectomy. To detect and analyse plaques from patients who underwent carotid endarterectomy over a period of time, to carry out follow-up, to monitor blood laboratory parameters, to perform data filtering, to analyse the type of plaque intracellular bacteria and the effect of different intracellular bacteria on postoperative adverse events, and to obtain the corresponding expected conclusions.

Secondary research objectives

1. to assess the species of intracellular bacteria in carotid plaques and to identify initially the relationship between intracellular bacteria and different cell species within the plaque;
2. to detect the correlation between the presence of intraplaque intracellular bacteria and the incidence of poor postoperative outcomes (cerebral infarction, carotid restenosis, and death), to identify the risk intracellular bacteria associated with poor outcomes, and to perform linear regression analyses to estimate the association between intracellular bacteria and plaque markers.
3. Information from clinical data was analysed, and regression analyses were performed to detect correlations between the presence of intracellular bacteria in risky plaques and the incidence of composite primary endpoints, corrected for age, sex, body mass index, total cholesterol, high-density lipoprotein and low-density lipoprotein cholesterol, triglycerides, creatinine, diabetes mellitus, hypertension, and previous cardiovascular events.

Overall design This study is a prospective, multicentre, cohort study. This registry study is expected to be conducted mainly at the Advanced Stroke Centre of Neurosurgery, Tang Du Hospital, with another 8-10 national advanced stroke centres participating in the study, with a study population of patients aged 18-80years undergoing CEA surgery. Patients who met all the inclusion criteria and did not fulfil any of the exclusion criteria could be considered for enrolment after indicating their informed consent to participate in this registry study and their willingness to sign an informed consent form.

All patients participating in this study underwent a comprehensive standardised assessment by a multidisciplinary team (including neurology, neurosurgery, haematology, endocrinology and other practitioners). The assessment included examination of neurology, neuropsychology and psychiatry, endocrine disorders, and haematological indices. Species identification of bacteria by bacterial 16SrDNA sequence sequencing will be performed and further verified by TEM, live bacterial staining methods.

The selected patients will receive routine surgical treatment and return for follow-up as recommended by the physician's follow-up, and the corresponding data generated from the clinical practice will be faithfully registered. Data and information generated by the clinical practice of patients will be recorded, including preoperative assessment, preoperative care, operating theatre care, anaesthesia management, intraoperative operation, postoperative medical management, postoperative care management and follow-up information.

Inclusion criteria

1. All patients were enrolled as first-time recipients of carotid endarterectomy;
2. site of lesion: beginning of internal carotid artery, bifurcation of internal and external carotid arteries;
3. symptomatic carotid stenosis with ≥70% stenosis on non-invasive examination or ≥50% stenosis on angiography;
4. patients with asymptomatic carotid stenosis with ≥70% stenosis on non-invasive examination or ≥60% stenosis on angiography;
5. asymptomatic carotid stenosis with non-invasive stenosis <70%, but angiographic or other evidence of unstable stenosis;
6. symptomatic carotid stenosis with a non-invasive stenosis of 50% to 69%;
7. sign an informed consent form.

Exclusion criteria

1. patients in poor general condition who do not tolerate general anaesthesia;
2. patients with psychiatric or severe psychological disorders;
3. patients with severe respiratory diseases
4. pregnant and lactating women;
5. patients who are participating in another clinical study
6. patients with advanced tumours or those who are expected to die within 1 year;

Study design protocol A. Methods: This study is a prospective, multicentre, cohort study. This registry study is expected to be conducted in the Department of Neurosurgery of Tang Du Hospital, and the target population of the study is adults aged 18-75 years old suffering from the need for carotid endarterectomy who are attending the Department of Neurosurgery of a tertiary general hospital. Patients who met all the inclusion criteria and did not meet any of the exclusion criteria could be considered for enrolment after indicating their informed consent to participate in this registry study and were willing to sign the informed consent form.

B. All patients participating in this study underwent a comprehensive standardised assessment by a multidisciplinary team (including neurology, neurosurgery, haematology, endocrinology and other practitioners). The assessment includes examination of neurology, neuropsychology and psychiatry, endocrine disorders, and haematological indices.

C. Selected patients will undergo routine surgical treatment and will be followed up by the practitioner's recommendations for follow-up, and the corresponding data generated by the clinical practice will be duly recorded. The data and information generated from the patients' clinical visits will be recorded, including preoperative assessment, preoperative care, operating theatre care, anaesthesia management, intraoperative operation, postoperative medical management, postoperative care management, and follow-up information.

D. Main items and contents of the experiment

1. assess the species of intracellular bacteria in carotid plaques, and initially identify the relationship between intracellular bacteria and different cell types within the plaque;
2. to detect the correlation between the presence of intracellular bacteria in plaques and the incidence of postoperative poor outcome (cerebral infarction, carotid restenosis, death), to identify the risk intracellular bacteria associated with poor outcome, and to perform linear regression analyses in order to estimate the associations between intracellular bacteria and plaque markers.
3. Information from clinical data was analysed, and regression analyses were performed to detect correlations between the presence of intracellular bacteria in risky plaques and the incidence of composite primary endpoints, corrected for age, sex, body mass index, total cholesterol, high-density lipoprotein and low-density lipoprotein cholesterol, triglycerides, creatinine, diabetes mellitus, hypertension, and previous cardiovascular events.

Information collection during the follow-up period Follow-up: Long-term post-discharge follow-up in the form of outpatient and telephone visits.

The follow-up visit includes: patient's general condition, including physical examination and necessary laboratory tests, necessary imaging tests and relevant scales, including the need for neuropsychiatric scoring. If a second operation or readmission occurs during the follow-up visit, it should be recorded accordingly. If additional laboratory tests are performed during follow-up, the original reports should be photocopied and filed in the patient's medical record. The patient's current medical history, hospitalisation, medication, especially the reason for change of medication, dosage, efficacy, and so on. The investigator is required to enter the laboratory test data into the eCRF (electronic Case Report Form) and keep the original laboratory report. The investigator should also provide the normal/abnormal judgement and the reference value range of the laboratory test data.

Timeframe of the study

The study will be divided into 2 phases as follows:

1. Preparation of the study: this phase encompasses the development of materials (CRF, EDC), informed consent form (Informed Consent Form (ICF), etc.), selection and evaluation of the study site, as well as the approval of the Ethics Committee, the development of the EDC system, the protocol and the initiation of the study site. This phase is expected to take 6 months;
2. Patient enrolment and completion of follow-up: estimated 30 months. The total duration of this study, from initiation to completion of the study summary report, is expected to be 36 months.

ELIGIBILITY:
Inclusion Criteria:

* All enrolled patients were diagnosed with clear head and neck artery stenosis and a risk event after head and neck revascularization;
* Location of lesion: origin of internal carotid artery, bifurcation of internal and external carotid arteries;
* Patients with symptomatic head and neck artery stenosis and dangerous events after head and neck blood flow reconstruction, and with a degree of stenosis ≥ 70% on non-invasive examination or stenosis ≥ 50% found on angiography;
* Asymptomatic head and neck artery stenosis and risk events after head and neck revascularization, with a degree of stenosis ≥ 70% on non-invasive examination or stenosis ≥ 60% found on angiography;
* Asymptomatic head and neck artery stenosis and dangerous events after head and neck blood flow reconstruction, with a non-invasive examination of stenosis degree less than 70%, but angiography or other examinations indicate that the stenosis lesion is in an unstable state;
* Symptomatic head and neck artery stenosis and risk events after head and neck revascularization, non-invasive examination of head and neck artery stenosis and risk event degree after head and neck revascularization at 50% to 69%

Exclusion Criteria:

* Patients with poor overall condition and intolerance to general anesthesia;
* Patients with mental illness or severe mental illness;
* Severe respiratory system diseases;
* Pregnant and lactating women;
* Participating in another clinical study;
* Patients with advanced tumors or those who are expected to die within one year;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a prospective, multicentre, cohort study. This registry study is expected to be conducted mainly at the Advanced Stroke Centre of Neurosurgery, Tang Du Hospital, with another 8-10 national advanced stroke centres participating in the study, with a study population of patients aged 18-80 years undergoing CEA surgery. Patients who met all the inclusion criteria and did not fulfil any of the exclusion criteria could be considered for enrolment after indicating their informed consent to participate in this registry study and their willingness to sign an informed consent form.
  All patients participating in this study underwent a comprehensive standardised assessment conducted by a multidisciplinary team. The assessment included examination of neurology, neuropsychology and psychiatry, endocrine disorders, and haematological indices. Species identification of bacteria by bacterial 16SrDNA sequence sequencing will be performed and further verified by TEM, live bacterial staining
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Types and distribution of intracellular bacteria in carotid plaques | 2023.01.01-2026.01.01
  Species identification of bacteria was carried out by sequencing of bacterial 16SrDNA sequences and further verified by TEM and live bacterial staining methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xian, Shanxi, China